CLINICAL TRIAL: NCT03551132
Title: Effects of Resistance Training Program on Physical Performance, Health Parameters and Quality of Life in Elderly (RTCHealth)
Brief Title: Effects of Resistance Training on Physical Performance, Health and Quality of Life in Elderly (RTCHealth)
Acronym: RTCHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Pablo Jorge Marcos Pardo, Principal investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UC PMAFI/03/12
Record Dates: First submitted 2018-05-15; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Sarcopenia; Body Weight Changes; Quality of Life
Keywords: elderly; resistance training; health
MeSH Terms: conditions — Sarcopenia; Body Weight Changes | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Experimental group A supervised progressive moderate-to-high RTC program designed to induce muscular hypertrophy was performed. EG followed a progressive moderate-to-high RTC program for 12-weeks. The training program incorporated resistance exercise of six major regions and consisted of 3 training sessions per week on non-consecutive days (Monday, Wednesday and Friday).
  All subjects performed the sets with moderate-intensity (8 to 12 repetitions) in each exercise and 30-60 seconds rest between sets. The load was increased during the 12 weeks from 60% 1-RM to high-intensity 80% 1-RM. The training load was increased when the individual could perform more than the prescribed number of repetitions (12 repetitions) followed the OMNI-RES scale and a hard effort perception level. Rest between sets was 1-2 minutes.
  Interventions: Other: Exercise test
- Group 2 (No Intervention): Control group The CG not participated in the RTC program.

INTERVENTIONS:
Other: Exercise test — Fat mass, Functional autonomy, muscular strength, quality of life questionnaire
  Arms: Group 1

SUMMARY:
Physical exercise is considered an important intervention for promoting well-being and healthy aging. The purpose of the present study was to determine the effects of moderate-to-high intensity resistance training circuit on different parameters of fat mass, functional autonomy, strength and quality of life in elderly. A randomized controlled trial was conducted. A total of 45 subjects, (27 females, 18 males) aged between 65-75 years old from Murcia (Spain) were randomly to experimental group (resistance training circuit for 12-weeks and isocaloric diet program) and control group (no resistance training intervention). Fat mass, functional autonomy, muscular strength, perceived exertion, and quality of life perception were obtained with validated tools. Experimental group decreases significantly their fat mass percentage whilst control group not presented differences. Muscular strength results exhibited significant differences between intervention training protocol. Furthermore, experimental group presented better marks than control group at quality of life questionnaire and functional autonomy scores. The moderate-to-high intensity resistance training circuit showed increase in upper and lower muscular strength as well as functional capacity and significantly decreased total fat mass and that improvements in physical function predict improvements in QoL perception in elderly.

DETAILED DESCRIPTION:
Participants and study design Figure 1 depicts a flowchart of this study. A total of 75 subjects were recruited from an elderly social groups and voluntarily participated in the study. After 9 subjects were excluded, 66 were ramdomly allocated to either the experimental group (EG, n= 33) or control group (CG, n= 33) at baseline. Subsequently, 25 subjects in the EG y 20 subjects in the CG completed the 12 weeks´follow-up assessments. The general characteristics of the subjects are given in Table 1. All subjects were originally from Murcia, Spain and were chosen according the following inclusion criteria: age ≥ 65 years, they never attended classes of fitness academies or following PA, and had no experience with ST. Exclusion criteria included any history of neuromuscular, metabolic, hormonal, cardiovascular diseases. Subjects were not taking any medication that could influence hormonal and neuromuscular metabolism. Participants were carefully informed about the possible risks and discomforts that could occur and were asked to complete a health history questionnaire and to sign a consent form. This study was performed in accordance with the standards of 1964 Declaration signed in Helsinki, and the protocol was approved by the Ethical Committee of the Catholic University of Murcia (UCAM), Spain.

Data collection pre and post-training (12 weeks) was performed in two days. On the first visit, between 8:00 and 9:00, biological test and quality of life measures were made. On the second day (24 hours after), the submaximal strength test was applied.

Nutrition and dietetics Isocaloric diets based on Mediterranean food were administrated at participants. Diets were analyzed and designed using Diet source software (Novartis, Barcelona, Spain), and were adapted accordingly to each particular subject. Diets were adjusted to strength exercises, including 1-1.2 g of protein/kg of body weight,36-38 25-30% of fat of total kcal and the remaining kcal was completed with carbohydrates as the main macronutrient, corresponding to 55-60% of total kcal. In general terms, the subjects performed 5 daily intakes. Daily energy intakes were adapted according to activity and frequency taking in account training and resting days.

Measures Fat mass Total body weight and % fat mass was measured after removal of shoes and heavy outer clothing, using a Tanita BC-418 MA (Tanita Corporation, Arlington Heights, IL) to the nearest 0.1 kg. Standing height without shoes was measured using a Seca 202 stadiometer (Seca, Hamburg, Germany) to the nearest 0.1 cm. BMI was calculated as the ratio of weight to squared height.

Functional autonomy The Latin American Group for Maturity (GDLAM) protocol was used to evaluate functional autonomy.15,40-42 It is composed of five tests: walking 10 m (W10m); standing up from a seated position (SSP); standing up from a prone position (SPP); standing up from a chair and moving about the room (SCMA); and putting on and taking off a shirt (PTS). These tests are used in a mathematical formula to calculate the GDLAM index (GI). The equipment used consisted of a 48-cm chair (measured from the seat to the floor), a stopwatch (Casio, Malaysia), two cones, a mat (Olive Fitness, Spain) and a sunny brand metal tape measure.

Muscular strength The predicted 1-repetition maximum (1-RM) testing protocol followed the procedure previously described by Brzycki. Upper body strength was measured by evaluating the strengths of the deltoids, triceps, and muscles by having the subjects perform a chest press (CHP) and military press (MP); lower body strength was measured by assessing the strengths of the gluteals, hamstrings, and quadriceps muscles by having them perform a leg extension (LE) and hip extension (HE). All machine based exercises were performed on Technogym equipment (Italy).

Perceived Exertion Ratings of perceived exertion were assessed using OMNI-RES scale of perceived exertion45,46 on an eleven-point scale (0= extremely easy to 10=extremely hard). Standard instructions for the OMNI-RES were read to the participants before each testing session. Previous evidence has supported the concurrent validity of this measure in performing upper and lower body resistance training programs.

Quality of life questionnaire Quality of Life in the elderly (WHOQOL-OLD)- a Spanish version: is an instrument developed by Power et al., translated and validated for the Spanish language. The WHOQOL-OLD is a 24-item self-report instrument that is divided into six Facets: Facet 1- Sensory Abilities (SA); Facet 2- Autonomy (A); Facet 3- Past, Present, and Future Activities (PPFA); Facet 4- Social Participation (SP); Facet 5- Death and Dying (DD); and Facet 6- Intimacy (I) (4 items per subscale). Each facet provides an individual score, and an overall score (general QoL - GQoL) is also calculated from the set of 24 items. Answers are based on a 5-point Likert response scale, with items 1, 2, 6, 7, 8, 9, 10 being reverse scored. Although all the response scales have five points they vary in their anchors: "Not at all"/ "An extreme amount"; "Completely"/ "Extremely"; "Very poor"/ "Very good"; "Very dissatisfied"/ "Very satisfied"; "Very unhappy"/ "Very happy"). Total scores on the WHOQOL-OLD range from 4 to 20, with higher scores being indicative of better quality of life (QoL).

All the test were administered in and indoor sports center, under the same environmental conditions for each participant.

Progressive moderate-to-high intensity RTC protocol Initially, prior to the commencement of the study, the subjects were submitted to two weeks of RTC, two sessions per week, in order to familiarize with the RTC exercises performed in the current study. During this familiarization period a higher emphasis was placed on learning the proper exercise techniques and brief pauses between repetitions were allowed in order to reset their starting positions when necessary48. In the second week, participants were also measured for body mass, height, fat mass, and quality of life questionnaires. In the same session, elderly completed the submaximal strength test 1-RM loads for chest press (CHP) and leg extension (LE), and the next day, completed the military press (MP), and hip extension (HE), and then, after 72 hours, the 1RM tests were repeated to determine test-retest reliability. In these testing sessions, participants were also familiarized with the OMNI-RES scale A supervised progressive moderate-to-high RTC program designed to induce muscular hypertrophy was performed. EG followed a progressive moderate-to-high RTC program for 12-weeks. The CG not participated in the RTC program. The training program incorporated resistance exercise of six major regions and consisted of 3 training sessions per week on non-consecutive days (Monday, Wednesday and Friday).

All subjects performed the sets with moderate-intensity (8 to 12 repetitions) in each exercise and 30-60 seconds rest between sets. The load was increased during the 12 weeks from 60% 1-RM to high-intensity 80% 1-RM. The training load was increased when the individual could perform more than the prescribed number of repetitions (12 repetitions) followed the OMNI-RES scale and a hard effort perception level. Rest between sets was 1-2 minutes.

All training sessions were monitored by a physical education professional expert and the subjects were not allowed to perform another exercises program during the training period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Never attended classes of fitness academies or following Physical Activity.
* No experience in Resistance Training.

Exclusion Criteria:

* No history of neuromuscular, metabolic, hormonal, cardiovascular diseases.
* Not taking any medication that could influence hormonal and neuromuscular metabolism.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
body weight in kilograms | Change from Baseline body weight (kg) at 12 weeks
  was measured after removal of shoes and heavy outer clothing, using a Tanita BC-418 MA (Tanita Corporation, Arlington Heights, IL) to the nearest 0.1 kg.
height in meters | Change from Baseline standing height (cm) at 12 weeks
  Standing height without shoes was measured using a Seca 202 stadiometer (Seca, Hamburg, Germany) to the nearest 0.1 cm.
Body Mass Index (BMI) | Change from Baseline Body Mass Index (BMI): (kg/m^2) at 12 weeks
  was calculated as the ratio of weight to squared height in kg/m^2
% Fat mass | Change from Baseline bioelectrical impedance % fat mass at 12 weeks
  % fat mass was measured after removal of shoes and heavy outer clothing, using a Tanita BC-418 MA (Tanita Corporation, Arlington Heights, IL) to the nearest 0.1 kg.
Quality of life | Change from Baseline Quality of Life perception at 12 weeks
  Quality of Life in the elderly (WHOQOL-OLD) is an instrument developed by Power et al., translated and validated for the Spanish language. The WHOQOL-OLD is a 24-item self-report instrument that is divided into six Facets. Is also calculated from the set of 24 items. Answers are based on a 5-point Likert response scale
Functional autonomy | Change from Baseline Functional autonomy at 12 weeks
  The Latin American Group for Maturity (GDLAM) protocol was used to evaluate functional autonomy. It is composed of five tests: W10m; SSP; SPP; SCMA; PTS. These tests are used in a mathematical formula to calculate the GDLAM index (GI).
Muscular strength | Change from Baseline Muscular Strength at 12 weeks
  The predicted 1-repetition maximum (1-RM) testing protocol followed the procedure previously described by Brzycki. Upper body muscles strength and lower body strength was measured

CONTACTS AND LOCATIONS:
Locations (1):
- Pablo Jorge Marcos Pardo, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No